CLINICAL TRIAL: NCT02867033
Title: National Clinical-biological Prospective Cohort of Incident Cases of Aggressive Fibromatosis
Brief Title: National Clinical-biological Prospective Cohort of Incident Cases of Aggressive Fibromatosis (ALTITUDES)
Acronym: ALTITUDES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Ligue contre le cancer, France (Other); Institut Curie (Other); Hôpital de la Timone (Other); SOS Desmoid e.V. (Unknown); APICIL funding (Unknown); GIRCI NO (Unknown); UNICANCER (Other); Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ALTITUDES-1508
Record Dates: First submitted 2016-07-15; First posted 2016-08-15 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Aggressive Fibromatosis
Keywords: desmoid tumour
MeSH Terms: conditions — Desmoid Tumors | interventions — Biopsy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study procedure (Other): Tumor biobank realization (biopsy...) and biobank constitution. coloscopy associated with colonic chromoscopy. Blood sampling (facultative). Pain evaluation
  Interventions: Procedure: biopsy; Other: biobank constitution; Procedure: Coloscopy; Procedure: Blood sampling (facultative); Other: Pain evaluation; Procedure: Tumor biobank realization

INTERVENTIONS:
Procedure: biopsy — pre-therapeutic or post-therapeutic biopsy or resected tissues
Other: biobank constitution — Constitution of a biobank with pre-therapeutic or post-therapeutic biopsy or resected tissues
Procedure: Coloscopy — For adult patients, a coloscopy with chromoscopy of ascending and sigmoid colon will be performed
Procedure: Blood sampling (facultative) — Blood sample can be collected at diagnostic or after medically significant events (progressive disease, local or systemic treatment, pregnancy...)
Other: Pain evaluation — Pain evaluation (EVA scale), anxiety (HADS questionnaire), quality of life questionnaire (EORTC-QLQ-C30)
Procedure: Tumor biobank realization — Realization of a tumor biobank is part of classical procedure of participating centers

SUMMARY:
The purpose of this study is to constitute the French largest Aggressive fibromatosis cohort.

DETAILED DESCRIPTION:
Aggressive fibromatosis (AF) is a rare non-metastasizing connective tissue tumor (< 300 cases/year in France), associated with high risk of local relapse, functional impairment and pain. AF can occur at any age, but most commonly between 25 and 40 with a significant female predominance. AF is most frequently (about 85%) sporadic and then associated with a somatic mutation of the CTNNB1 gene. AF is associated with heredity condition, as complication of familial adenomatous polyposis (with germinal mutation of Adenomatous polyposis coli (APC) gene). Most of AF arises on lims or abdominal wall. Nevertheless, some particular locations are life-threatening (mesenteric or cervical locations). The natural course of AF is unpredictable. One third of tumors are spontaneously stable. One third of tumor spontaneously decreases. One third of tumor is progressive, with a non-linear tumor growth dynamic. As the consequence the decision making for starting curative intent treatment is difficult, since some treatment could be mutilating (large en bloc surgery) or associated with late and severe complications (radiotherapy) and since these treatments could fail to control this benign tumor. Therapeutic options are: wait-and-see policy, surgery (sometimes mutilating), radiotherapy or systemic treatment (non-steroidal anti-inflammatory drugs, hormonotherapy, imatinib, chemotherapy). Level of evidence associated these options is very low, based on retrospective studies and rare non-randomized phase II clinical trials.

Regarding these uncertainties, physicians can hardly answer to patient questions.

Prospective data provided by a large multi-center cohort is needed. The objective of the present study is to create a large cohort of incident cases of AF associated with tumor bank and collection of blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Incident Case of aggressive fibromatosis in France, diagnosed after 01/01/2016
* Confirmed diagnosis by the French anatomopathological diagnosis network (including search for mutation of the β-Catenin Gene, CTNNB1)
* Affiliation to the National Health System
* Informed consent signed (both parents signature for non adult patients)

Exclusion Criteria:

* Administrative or legal measure of liberty privation
* Patient not able to give consent or unwilling to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Incident cases of aggressive fibromatosis, diagnosed after 01/01/2016 in France | through study completion, an average of 5 years
  To constitute, at a national level, the largest cohort of incident cases of desmoid tumours

SECONDARY OUTCOMES:
Number of Aggressive Fibromatosis associated with familial adenomatous polyposis | through study completion, an average of 5 years
  To describe and analyse the link between Aggressive Fibromatosis and familial adenomatous polyposis
Percentage of CTNNB1 mutation in non-selected cases of Aggressive Fibromatosis | through study completion, an average of 5 years
  To describe the proportion of AF cases characterized by CTNNB1 somatic mutation
Management of AF | through study completion, an average of 5 years
  Description of the management of AF. Study of prognosis factor for progressive disease and death. Study of tumor response to treatments (Best response and progression-free survival) according to RECIST 1.1.
Hospital Anxiety and Depression Scale (HADS) | at baseline, one year
  To describe the psychological impact of the disease at diagnosis and a year after diagnosis. And to compare changes between the time of diagnosis and one year after the treatments used.
Quality of Life Questionnaire (QLQC30) | at baseline, one year
  To describe the consequences of the disease on the quality of life at diagnosis and a year after diagnosis. And to compare changes between the time of diagnosis and one year after the treatments used.
Impact of pregnancy and hormonal exposure | Through study completion, an average of 5 years
  To study the impact of pregnancy and hormonal exposure on the evolution of the disease according to recurrence/progression rates
Incidence of polyposis and colorectal cancer | Through study completion, an average of 5 years
  Rate of polyposis and colorectal cancer in the AF population

OTHER OUTCOMES:
Mutation rate of APC | through study completion, an average of 5 years
  To determine the mutation rate of APC at constitutional and somatic levels
Mutation rate of CTNNB1 | through study completion, an average of 5 years
  To determine the mutation rate of CTNNB1 at constitutional and somatic levels
Correlation between APC and CTNNB1 mutations rates | through study completion, an average of 5 years
  To demonstrate that APC and CTNNB1 mutations are two mutually exclusive molecular alterations
APC mutation rate | through study completion, an average of 5 years
  To correlate mutational somatic and constitutional rate of APC gene
Occurrence of other mutations | through study completion, an average of 5 years
  To search other molecular anomalies for patients without APC or CTNNB1 mutations (10 % of cases)
Cell free (circulating) nucleic acid extraction technics | through study completion, an average of 5 years
  To determine sensibility and specificity of cell free (circulating) nucleic acid extraction techniques
AF outcome | through study completion, an average of 5 years
  To describe patient outcomes and identify prognostic factors
Treatment response | through study completion, an average of 5 years
  To search for factors involved in response treatment prediction

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, PhD, Principal Investigator — Centre Oscar Lambret; Sébastien SALAS, PhD, Principal Investigator — Hopital Timone adultes
Locations (39):
- France (39):
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - CHU Angers, Angers
  - CHU de Besançon, Besançon
  - Hôpital des Enfants, Bordeaux
  - Institut Bergonié, Bordeaux
  - CHU de Caen-Côte de Nacre, Caen
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - CHU de Grenoble- Hôpital Couple Enfant, Grenoble
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Hôpital la Timone Enfants Service Oncologie Pédiatrique, Marseille
  - Hôpital la Timone Service Oncologie Médicale, Marseille
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Hôpital Mère Enfant - CHU Nantes, Nantes
  - Hôpital Archet 2, Nice
  - Institut Curie Département Oncologie Médicale, Paris
  - Institut Curie Département Oncologie Pédiatrique, Paris
  - Hôpital Saint Louis, Paris
  - Hôpîtal d'Enfants Armand Trousseau, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint Antoine, Paris
  - CHU de Reims, Reims
  - CHU de Rennes- Hôpital Sud, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie-Hôpital René Huguenin, Saint-Cloud
  - CHU Saint-Étienne - Hôpital Nord, Saint-Etienne
  - Hôpital Privé de la Loire, Saint-Etienne
  - Institut de Cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - Institut de Cancérologie et d'Hématologie Universitaire de Saint Etienne, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CHU Toulouse - Hôpital des Enfants, Toulouse
  - Institut Claudius Régaud, Toulouse
  - CHU Tours - Clocheville, Tours
  - Hôpital d'Enfants- CHU Nancy, Vandœuvre-lès-Nancy
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Penel N, Bonvalot S, Bimbai AM, Meurgey A, Le Loarer F, Salas S, Piperno-Neumann S, Chevreau C, Boudou-Rouquette P, Dubray-Longeras P, Kurtz JE, Guillemet C, Bompas E, Italiano A, Le Cesne A, Orbach D, Thery J, Le Deley MC, Blay JY, Mir O. Lack of Prognostic Value of CTNNB1 Mutation Profile in Desmoid-Type Fibromatosis. Clin Cancer Res. 2022 Sep 15;28(18):4105-4111. doi: 10.1158/1078-0432.CCR-21-4235. PMID 35294527